CLINICAL TRIAL: NCT02064816
Title: Multicenter, Open-label, 12 Week, Phase IV Prospective Randomized Study Aimed at Evaluating Whether sc IFN Beta 1a (Rebif®) Administered in the Morning May Affect the Severity of Flu-like Syndrome and Patient-perceived Invisible Symptoms in Subjects With Relapsing Multiple Sclerosis
Brief Title: A Study of Rebif® in Subjects With Relapsing Multiple Sclerosis
Acronym: RELIEF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200136-570; 2013-004450-21 (EudraCT Number)
Record Dates: First submitted 2014-02-13; First posted 2014-02-17 (Estimated); Results first posted 2018-09-20 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-01

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis, Relapsing-Remitting; Interferon beta 1a; Rebif®
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1a

ARMS (2):
- Rebif® Morning Administration (Experimental)
  Interventions: Drug: Rebif®
- Rebif® Evening Administration (Experimental)
  Interventions: Drug: Rebif®

INTERVENTIONS:
Drug: Rebif® — Rebif® will be administered at a dose of 44 microgram (mcg) subcutaneously three times a week in the morning using RebiSmart® self-injector device for 12 weeks.
  Arms: Rebif® Morning Administration
Drug: Rebif® — Rebif® will be administered at a dose of 44 mcg subcutaneously three times a week in the evening using RebiSmart® self-injector device for 12 weeks.
  Arms: Rebif® Evening Administration

SUMMARY:
This is an open-label, multi-center, 12-week, randomized, controlled, parallel group, Phase 4 study to assess whether the morning administration of interferon beta 1a (Rebif®) leads to a lower severity of flu-like symptoms (FLS) as compared to the evening administration, in subjects with relapsing multiple sclerosis (RMS).

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 60 years of age
* Female subjects must be neither pregnant nor breast-feeding and must lack child-bearing potential. Furthermore, female subjects must not have been pregnant from at least three months prior to enter in the study
* Subjects have RMS according to the revised McDonald Criteria (2010)
* Subjects with an expanded disability status scale (EDSS) score of less than 6.0
* Subjects naive to treatment and eligible for treatment with Rebif® 44 three times a week, or patients having received glatiramer acetate with a wash-out from at least one month, or patients having received treatment with natalizumab or fingolimod with a wash-out from at least three months
* Subjects able to self-inject treatment using RebiSmart®
* Subjects willing and able to comply with the protocol for the duration of the study
* Subjects have given written informed consent to take part in the study

Exclusion Criteria:

* Subjects have any disease other than MS that could better explain his/her signs and symptoms
* Subjects who have received any immunosuppressive agents within 3 months prior to Baseline
* Subjects who have received any corticosteroids within 30 days prior to Baseline
* Subjects have a MS relapse within 30 days prior to Baseline
* Subjects have inadequate liver function and bone marrow reserve as defined in the protocol
* Subjects have moderate to severe renal impairment
* Subjects have any visual or physical impairment that precludes the subjects from self-injecting the treatment using RebiSmart®
* Subjects have hypersensitivity to natural or recombinant interferon, or to any of its excipients
* Subjects have any contra-indications to treatment with interferon (IFN) beta 1a according to Summary of Product Characteristics (SmPC)
* Subjects have any contra-indications to treatment with ibuprofen/paracetamol according to SmPC
* Obese subjects, defined by body mass index greater than 30 kilogram per square meter (kg/m^2)
* Subjects have participated in any other investigational trial within 30 days from Baseline
* Subjects have any other significant disease that in the Investigator's opinion would exclude the subject from the trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2014-05-31 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono S.P.A., Italy
Locations (1):
- Please contact the Merck KGaA Communication Center, Darmstadt, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 29 clinical trial sites in Italy.
Pre-assignment Details: A total of 200 subjects were enrolled in the study, of which 104 were randomized to Rebif morning treatment group, and 96 were randomized to Rebif evening treatment group. A subgroup of subjects also took part in a sub study assessing cytokines and other immunological biomarkers.
Groups:
- Rebif Morning Administration: Subjects self-injected Rebif at a dose of 44 microgram (mcg) subcutaneously three times a week by using RebiSmart autoinjector device in the morning for 12 weeks.
- Rebif Evening Administration: Subjects self-injected Rebif at a dose of 44 mcg subcutaneously three times a week by using RebiSmart autoinjector device in the evening for 12 weeks.
Period: Overall Study
Arm/Group | Rebif Morning Administration | Rebif Evening Administration
Started | 104 | 96
Completed | 96 | 88
Not Completed | 8 | 8
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Therapeutic failure | 0 | 1
Not completed — Other | 1 | 3

BASELINE CHARACTERISTICS:
Population: The Intention to Treat Analysis Set (ITT) included all subjects enrolled into the study and assigned to the RebiSmart device.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rebif Morning Administration | Rebif Evening Administration | Total
Number analyzed (Participants) | 104 | 96 | 200
Age, Customized [Number; unit: subjects]
  <18 years | 0 | 0 | 0
  >=18 years to 64 years | 104 | 96 | 200
  >64 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 62 | 138
  Male | 28 | 34 | 62

OUTCOME MEASURES:

1. Primary Outcome: Difference in Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Flu Like Symptom (FLS) Score Between Rebif Morning Administration and Rebif Evening Administration Groups at Week 12
Description: The MSTCQ was used as a tool to measure treatment satisfaction, focusing on the attributes specific to multiple sclerosis (MS) medications. The FLS subscale of MSTCQ was defined as the sum of the scores for questions 13 to 16 with a minimum possible total FLS score = 1 and a maximum possible total FLS score = 20. Lower score indicates lower flu like symptoms and better satisfaction. Difference between Rebif Morning Administration and Rebif Evening Administration groups at Week 12 is presented in statistical analysis section.
Time Frame: Week 12
Population: The ITT included all subjects enrolled into the study and assigned to the RebiSmart device. Here, "Number of Subjects Analyzed" signifies those subjects who were evaluable for this outcome measure. Missing data on FLS were imputed using the last observation carried forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Rebif Morning Administration | Rebif Evening Administration
Number analyzed (Participants) | 99 | 88
units on scale | 12.3 (3.87) | 11.8 (3.02)
Statistical Analysis 1: Comparison: Rebif Morning Administration vs Rebif Evening Administration; Test type: Superiority or Other; p = 0.277763, Mann-Whitney Non Parametric test; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.46 to 1.56], Standard Deviation 3.50

2. Secondary Outcome: Difference in Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Flu Like Symptom (FLS) Score Between Rebif Morning Administration and Rebif Evening Administration Groups at Week 4 and 8
Description: The MSTCQ was used as a tool to measure treatment satisfaction, focusing on the attributes specific to multiple sclerosis (MS) medications. The FLS subscale of MSTCQ was defined as the sum of the scores for questions 13 to 16 with a minimum possible total FLS score = 1 and a maximum possible total FLS score = 20. Lower score indicates lower flu like symptoms and better satisfaction. Difference between Rebif Morning Administration and Rebif Evening Administration groups at Week 4 and 8 is presented in statistical analysis section.
Time Frame: Week 4 and 8
Population: The ITT included all subjects enrolled into the study and assigned to the RebiSmart device. Here, "Number of Subjects Analyzed" signifies those subjects who were evaluable for this outcome measure. Here "Number Analyzed" signifies those subjects who were evaluable for this outcome measure for specified category.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Rebif Morning Administration | Rebif Evening Administration
Number analyzed (Participants) | 99 | 88
units on scale
  Week 4: number analyzed (Participants) | 81 | 81
  Week 4 | 12.4368 [11.7402 to 13.1333] | 11.0876 [10.3705 to 11.8046]
  Week 8: number analyzed (Participants) | 97 | 88
  Week 8 | 13.0039 [12.3244 to 13.6834] | 11.6672 [10.9565 to 12.3779]
Statistical Analysis 1: Comparison: Rebif Morning Administration vs Rebif Evening Administration; Week 4; Test type: Superiority or Other; p = 0.0083, linear mixed model for repeated measures; Least Square (LS) Mean difference = 1.3492, 95% CI 2-sided [0.3495 to 2.3489]
Statistical Analysis 2: Comparison: Rebif Morning Administration vs Rebif Evening Administration; Week 8; Test type: Superiority or Other; p = 0.0079, linear mixed model for repeated measures; LS Mean difference = 1.3367, 95% CI 2-sided [0.3534 to 2.3200]

3. Secondary Outcome: Difference in Multiple Sclerosis Treatment Concern Questionnaire (MSTCQ) Subscale Scores Between Rebif Morning Administration and Rebif Evening Administration Groups at Week 4, 8 and 12
Description: MSTCQ was used as a tool to measure treatment satisfaction, focusing on attributes specific to MS medications. Following sub-scales were assessed: Injection site reactions (ISRs), Global side-effects, Benefits, Pain, Visual Analog Scale (VAS), and Rating of Pain. ISR subscale was defined as sum of scores for questions 17 to 20, with a minimum possible total score of 4 and a maximum possible total score of 20. Global side-effects subscale was defined as sum of scores for questions 21 to 23 with minimum possible total score of 3 and a maximum possible total score of 15. Benefits (question 35); description of pain (question 36); VAS (question 37); rating of pain (question 38) subscales ranged from minimum possible score of 1 and a maximum possible total score of 5. For each of the subscales, lower scores indicated better satisfaction. Difference between both the groups at Week 4, 8 and 12 for individual sub-scales is presented in statistical analysis section.
Time Frame: Week 4, 8 and 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Rebif Morning Administration | Rebif Evening Administration
Number analyzed (Participants) | 103 | 93
units on scale
  ISRs subscale Week 4: number analyzed (Participants) | 75 | 66
  ISRs subscale Week 4 | 10.8459 [10.1609 to 11.5309] | 10.4456 [9.7177 to 11.1735]
  ISRs subscale Week 8: number analyzed (Participants) | 80 | 77
  ISRs subscale Week 8 | 11.5363 [10.8625 to 12.2101] | 11.4515 [10.7540 to 12.1490]
  ISRs subscale Week 12: number analyzed (Participants) | 83 | 75
  ISRs subscale Week 12 | 11.6380 [10.9720 to 12.3041] | 11.9625 [11.2598 to 12.6652]
  Global side-effect subscale: Week 4: number analyzed (Participants) | 96 | 91
  Global side-effect subscale: Week 4 | 10.2144 [9.6771 to 10.7518] | 10.2852 [9.7276 to 10.8429]
  Global side-effect subscale: Week 8: number analyzed (Participants) | 94 | 87
  Global side-effect subscale: Week 8 | 10.4111 [9.8698 to 10.9525] | 10.2214 [9.6567 to 10.7862]
  Global side-effect subscale: Week 12: number analyzed (Participants) | 93 | 87
  Global side-effect subscale: Week 12 | 10.5879 [10.0456 to 11.1302] | 10.1782 [9.6132 to 10.7432]
  Benefits: Week 4: number analyzed (Participants) | 76 | 75
  Benefits: Week 4 | 3.1325 [2.7856 to 3.4794] | 3.5408 [3.1912 to 3.8905]
  Benefits: Week 8: number analyzed (Participants) | 71 | 74
  Benefits: Week 8 | 3.5779 [3.2207 to 3.9351] | 3.7137 [3.3622 to 4.0652]
  Benefits: Week 12: number analyzed (Participants) | 70 | 71
  Benefits: Week 12 | 3.6059 [3.2467 to 3.9652] | 3.6640 [3.3062 to 4.0218]
  Description of pain: Week 4: number analyzed (Participants) | 89 | 86
  Description of pain: Week 4 | 4.3755 [3.2024 to 5.5485] | 3.7846 [2.5846 to 4.9847]
  Description of pain: Week 8: number analyzed (Participants) | 85 | 84
  Description of pain: Week 8 | 5.3132 [4.1262 to 6.5003] | 6.0821 [4.8767 to 7.2875]
  Description of pain: Week 12: number analyzed (Participants) | 88 | 80
  Description of pain: Week 12 | 5.7853 [4.6089 to 6.9617] | 5.6431 [4.4239 to 6.8624]
  VAS: Week 4: number analyzed (Participants) | 96 | 89
  VAS: Week 4 | 11.8837 [7.6691 to 16.0983] | 11.2293 [6.8280 to 15.6305]
  VAS: Week 8: number analyzed (Participants) | 91 | 87
  VAS: Week 8 | 17.2316 [12.9597 to 21.5035] | 19.4610 [15.0359 to 23.8860]
  VAS: Week 12: number analyzed (Participants) | 91 | 84
  VAS: Week 12 | 16.1757 [11.9054 to 20.4460] | 21.5953 [17.1359 to 26.0547]
  Rating of pain: Week 4: number analyzed (Participants) | 98 | 90
  Rating of pain: Week 4 | 1.3073 [1.1008 to 1.5138] | 1.3004 [1.0846 to 1.5162]
  Rating of pain: Week 8: number analyzed (Participants) | 93 | 89
  Rating of pain: Week 8 | 1.5653 [1.3553 to 1.7753] | 1.6522 [1.4356 to 1.8688]
  Rating of pain: Week 12: number analyzed (Participants) | 93 | 86
  Rating of pain: Week 12 | 1.4994 [1.2895 to 1.7094] | 1.7218 [1.5029 to 1.9407]
Statistical Analysis 1: Comparison: Rebif Morning Administration vs Rebif Evening Administration; ISRs subscale Week 4; Test type: Superiority or Other; p = 0.4311, linear mixed model for repeated measures; LS Mean difference = 0.4003, 95% CI 2-sided [-0.5992 to 1.3998]
Statistical Analysis 2: Comparison: Rebif Morning Administration vs Rebif Evening Administration; ISRs subscale Week 8; Test type: Superiority or Other; p = 0.8635, linear mixed model for repeated measures; LS Mean difference = 0.08479, 95% CI 2-sided [-0.8850 to 1.0546]
Statistical Analysis 3: Comparison: Rebif Morning Administration vs Rebif Evening Administration; ISRs subscale Week 12; Test type: Superiority or Other; p = 0.5099, linear mixed model for repeated measures; LS Mean difference = -0.3245, 95% CI 2-sided [-1.2927 to 0.6437]
Statistical Analysis 4: Comparison: Rebif Morning Administration vs Rebif Evening Administration; Global side-effect subscale: Week 4; Test type: Superiority or Other; p = 0.8574, linear mixed model for repeated measures; LS Mean difference = -0.07079, 95% CI 2-sided [-0.8452 to 0.7036]
Statistical Analysis 5: Comparison: Rebif Morning Administration vs Rebif Evening Administration; Global side-effect subscale: Week 8; Test type: Superiority or Other; p = 0.6338, linear mixed model for repeated measures; LS Mean difference = 0.1897, 95% CI 2-sided [-0.5926 to 0.9720]
Statistical Analysis 6: Comparison: Rebif Morning Administration vs Rebif Evening Administration; Global side-effect subscale: Week 12; Test type: Superiority or Other; p = 0.3042, linear mixed model for repeated measures; LS Mean difference = 0.4097, 95% CI 2-sided [-0.3734 to 1.1929]
Statistical Analysis 7: Comparison: Rebif Morning Administration vs Rebif Evening Administration; Benefits: Week 4; Test type: Superiority or Other; p = 0.1038, linear mixed model for repeated measures; LS Mean difference = -0.4083, 95% CI 2-sided [-0.9008 to 0.08419]
Statistical Analysis 8: Comparison: Rebif Morning Administration vs Rebif Evening Administration; Benefits: Week 8; Test type: Superiority or Other; p = 0.5940, linear mixed model for repeated measures; LS Mean difference = -0.1358, 95% CI 2-sided [-0.6370 to 0.3653]
Statistical Analysis 9: Comparison: Rebif Morning Administration vs Rebif Evening Administration; Benefits: Week 12; Test type: Superiority or Other; p = 0.8217, linear mixed model for repeated measures; LS Mean difference = -0.05809, 95% CI 2-sided [-0.5651 to 0.4489]
Statistical Analysis 10: Comparison: Rebif Morning Administration vs Rebif Evening Administration; Description of pain: Week 4; Test type: Superiority or Other; p = 0.4890, linear mixed model for repeated measures; LS Mean difference = 0.5909, 95% CI 2-sided [-1.0873 to 2.2690]
Statistical Analysis 11: Comparison: Rebif Morning Administration vs Rebif Evening Administration; Description of pain: Week 8; Test type: Superiority or Other; p = 0.3719, linear mixed model for repeated measures; LS Mean difference = -0.7689, 95% CI 2-sided [-2.4607 to 0.9229]
Statistical Analysis 12: Comparison: Rebif Morning Administration vs Rebif Evening Administration; Description of pain: Week 12; Test type: Superiority or Other; p = 0.8690, linear mixed model for repeated measures; LS Mean difference = 0.1422, 95% CI 2-sided [-1.5521 to 1.8364]
Statistical Analysis 13: Comparison: Rebif Morning Administration vs Rebif Evening Administration; VAS: Week 4; Test type: Superiority or Other; p = 0.8328, linear mixed model for repeated measures; LS Mean difference = 0.6544, 95% CI 2-sided [-5.4393 to 6.7482]
Statistical Analysis 14: Comparison: Rebif Morning Administration vs Rebif Evening Administration; VAS: Week 8; Test type: Superiority or Other; p = 0.4764, linear mixed model for repeated measures; LS Mean difference = -2.2294, 95% CI 2-sided [-8.3800 to 3.9212]
Statistical Analysis 15: Comparison: Rebif Morning Administration vs Rebif Evening Administration; VAS: Week 12; Test type: Superiority or Other; p = 0.0852, linear mixed model for repeated measures; LS Mean difference = -5.4196, 95% CI 2-sided [-11.5939 to 0.7547]
Statistical Analysis 16: Comparison: Rebif Morning Administration vs Rebif Evening Administration; Rating of pain: Week 4; Test type: Superiority or Other; p = 0.9639, linear mixed model for repeated measures; LS Mean difference = 0.006873, 95% CI 2-sided [-0.2918 to 0.3055]
Statistical Analysis 17: Comparison: Rebif Morning Administration vs Rebif Evening Administration; Rating of pain: Week 8; Test type: Superiority or Other; p = 0.5715, linear mixed model for repeated measures; LS Mean difference = -0.08689, 95% CI 2-sided [-0.3886 to 0.2148]
Statistical Analysis 18: Comparison: Rebif Morning Administration vs Rebif Evening Administration; Rating of pain: Week 12; Test type: Superiority or Other; p = 0.1502, linear mixed model for repeated measures; LS Mean difference = -0.2224, 95% CI 2-sided [-0.5256 to 0.08090]

4. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) Score at Week 4, 8 and 12
Description: HADS was used to measure depression and anxiety in subjects. The scale was limited to 14 questions. Seven of the items related to anxiety and 7 related to depression. Each item on the questionnaire was scored from 0-3 giving a total score between 0 and 21 for either anxiety or depression where higher score indicates more anxiety/depression.
Time Frame: Baseline, Week 4, 8 and 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Rebif Morning Administration | Rebif Evening Administration
Number analyzed (Participants) | 101 | 93
units on scale
  Anxiety score: Change at Week 4: number analyzed (Participants) | 95 | 90
  Anxiety score: Change at Week 4 | -0.6625 [-1.1976 to -0.1273] | -0.4604 [-1.0106 to 0.08968]
  Anxiety score: Change at Week 8: number analyzed (Participants) | 89 | 88
  Anxiety score: Change at Week 8 | -0.7222 [-1.2688 to -0.1755] | -0.3763 [-0.9308 to 0.1782]
  Anxiety score: Change at Week 12: number analyzed (Participants) | 90 | 86
  Anxiety score: Change at Week 12 | -0.6435 [-1.1879 to -0.09918] | 0.05023 [-0.5081 to 0.6085]
  Depression score: Change at Week 4: number analyzed (Participants) | 97 | 89
  Depression score: Change at Week 4 | -0.1539 [-0.8083 to 0.5005] | 0.2211 [-0.4617 to 0.9038]
  Depression score: Change at Week 8: number analyzed (Participants) | 92 | 89
  Depression score: Change at Week 8 | -0.2397 [-0.9062 to 0.4267] | 0.1999 [-0.4835 to 0.8833]
  Depression score: Change at Week 12: number analyzed (Participants) | 91 | 86
  Depression score: Change at Week 12 | 0.1906 [-0.4778 to 0.8590] | 0.1162 [-0.5741 to 0.8066]

5. Secondary Outcome: Change From Baseline in Fatigue Severity Scale (FSS) Score at Week 4, 8 and 12
Description: FSS is a method designed to assess disabling fatigue in all the individuals. The Fatigue Severity Scale is a 9-item questionnaire developed to assess the level of fatigue due to neurological disease, were each item assessed on a 1-7 scale (1= no fatigue and 7= severe fatigue). The total score was calculated as the average of individual 9-items and ranged from 1 to 7 with a higher value indicating greater impairment due to fatigue.
Time Frame: Baseline, Week 4, 8 and 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Rebif Morning Administration | Rebif Evening Administration
Number analyzed (Participants) | 98 | 94
units on scale
  Change at Week 4: number analyzed (Participants) | 93 | 92
  Change at Week 4 | 0.2089 [-0.05810 to 0.4759] | 0.06901 [-0.2010 to 0.3391]
  Change at Week 8: number analyzed (Participants) | 92 | 90
  Change at Week 8 | 0.2062 [-0.06211 to 0.4746] | 0.1366 [-0.1354 to 0.4085]
  Change at Week 12: number analyzed (Participants) | 88 | 87
  Change at Week 12 | 0.1464 [-0.1253 to 0.4182] | 0.1942 [-0.08036 to 0.4688]

6. Secondary Outcome: Change From Baseline in Pittsburgh Sleep Quality Index (PSQI) Score at Week 4, 8 and 12
Description: PSQI is a self-rated questionnaire which assess sleep quality and disturbances over a 1-month interval using seven clinically derived components of sleep difficulties: sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction. PSQI is a summary of 7 components. Each component is scored from 0 to 3, therefore PSQI has a range of 0 (better) to 21 (worse). Interpretation of the PSQI is that a score less than 5 is associated with good sleep quality and a score of 5 or greater is associated with poor sleep quality.
Time Frame: Baseline, Week 4, 8 and 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Rebif Morning Administration | Rebif Evening Administration
Number analyzed (Participants) | 69 | 55
units on scale
  Change at Week 4: number analyzed (Participants) | 58 | 50
  Change at Week 4 | -0.08889 [-0.7690 to 0.5912] | 0.5747 [-0.1653 to 1.3147]
  Change at Week 8: number analyzed (Participants) | 62 | 53
  Change at Week 8 | -0.4513 [-1.1161 to 0.2136] | 0.7092 [-0.01588 to 1.4343]
  Change at Week 12: number analyzed (Participants) | 53 | 47
  Change at Week 12 | 0.07841 [-0.6265 to 0.7833] | 0.4293 [-0.3270 to 1.1855]

7. Secondary Outcome: Change From Baseline in Multiple Sclerosis International Quality of Life (MusiQOL) Score at Week 4, 8 and 12
Description: The MusiQoL is a validated 31-item questionnaire describing 9 dimensions: activities of daily living (8 items); psychological well-being (4 items); symptoms (3 items); relationships with friends (4 items); relationships with family (3 items); relationship with healthcare system (3 items); sentimental and sexual life (2 items); coping (2 items); and rejection (2 items). Each of the questions was answered using a 6-point Likert scale ranging from 1 (never/not at all) to 6 (always/very much). The scores of each dimension were obtained by computing mean of the item scores of dimension with negatively worded item scores reversed so that higher scores indicated higher health-related quality of life (QoL). All 9 dimension scores were linearly transformed to a 0 to 100 scale and the average of the 9 dimensions was used to give a Global Score ranging from 0 to 100, where higher scores indicated higher health-related quality of life (QoL).
Time Frame: Baseline, Week 4, 8 and 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Rebif Morning Administration | Rebif Evening Administration
Number analyzed (Participants) | 89 | 85
units on scale
  Global Score: Change at Week 4: number analyzed (Participants) | 83 | 81
  Global Score: Change at Week 4 | 1.6283 [-0.3761 to 3.6326] | 0.1174 [-1.9196 to 2.1544]
  Global Score: Change at Week 8: number analyzed (Participants) | 81 | 78
  Global Score: Change at Week 8 | 1.1439 [-0.8780 to 3.1658] | -2.2945 [-4.3568 to -0.2321]
  Global Score: Change at Week 12: number analyzed (Participants) | 78 | 75
  Global Score: Change at Week 12 | 0.9670 [-1.0753 to 3.0094] | -1.3948 [-3.4796 to 0.6900]

8. Secondary Outcome: Percentage of Subjects With Treatment Adherence at Week 4, 8 and 12
Description: Adherence to treatment was calculated as 100 x the number of completed injections the subject administered divided by the expected number of injections. Treatment adherence was divided in two categories: percentage of subjects with less than (<) 80 percent adherence and percentage of subjects with more than or equal to (>=) 80 percent adherence.
Time Frame: Week 4, 8 and 12
Population: as for outcome 2
Measure: Number; unit: Percentage of subjects
Arm/Group | Rebif Morning Administration | Rebif Evening Administration
Number analyzed (Participants) | 92 | 85
Percentage of subjects
  < 80 percent adherence at Week 4 | 3.3 | 5.9
  >= 80 percent adherence at Week 4 | 96.7 | 94.1
  < 80 percent adherence at Week 8: number analyzed (Participants) | 69 | 67
  < 80 percent adherence at Week 8 | 2.9 | 1.5
  >= 80 percent adherence at Week 8: number analyzed (Participants) | 69 | 67
  >= 80 percent adherence at Week 8 | 97.1 | 98.5
  < 80 percent adherence at Week 12: number analyzed (Participants) | 84 | 79
  < 80 percent adherence at Week 12 | 4.8 | 6.3
  >= 80 percent adherence at Week 12: number analyzed (Participants) | 84 | 79
  >= 80 percent adherence at Week 12 | 95.2 | 93.7

9. Secondary Outcome: Change From Baseline in Circulating Levels of Cytokines at Week 12
Description: Results are presented for three cytokines: leptin, resistin and adiponectin.
Time Frame: Baseline and Week 12
Population: The ITT included all subjects enrolled into the study and assigned to the RebiSmart device. Here, "Number of Subjects Analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: microgram per liter (mcg/L)
Arm/Group | Rebif Morning Administration | Rebif Evening Administration
Number analyzed (Participants) | 89 | 77
microgram per liter (mcg/L)
  Leptin: Change at Week 12 | -2.6 (3.42) | -2.6 (3.90)
  Resistin: Change at Week 12 | -3.1 (3.31) | -3.0 (3.77)
  Adiponectin: Change at Week 12 | 2.8 (6.38) | 2.8 (5.51)

10. Secondary Outcome: Correlation Between Change From Baseline in Circulating Levels of Cytokines (Leptin, Resistin and Adiponectin) and in Flu Like Symptom (FLS) Score at Week 12
Description: Correlation was assessed by using Pearson correlation coefficient. The MSTCQ was used as a tool to measure treatment satisfaction, focusing on the attributes specific to MS medications. The FLS subscale of MSTCQ was defined as the sum of the scores for questions 13 to 16 with a minimum possible total FLS score = 1 and a maximum possible total FLS score = 20. Lower score indicates lower flu like symptoms and better satisfaction.
Time Frame: Baseline and Week 12
Population: as for outcome 9
Measure: Number; unit: Correlation coefficient
Arm/Group | Rebif Morning Administration | Rebif Evening Administration
Number analyzed (Participants) | 77 | 70
Correlation coefficient
  Leptin and FLS: Change at Week 12 | 0.08822 | 0.03944
  Resistin and FLS: Change at Week 12 | -0.20200 | -0.01069
  Adiponectin and FLS: Change at Week 12 | 0.04616 | -0.13571

11. Secondary Outcome: Correlation Between Change From Baseline in Circulating Levels of Cytokines and in Other MSTCQ Items, HADS, FSS, PSQI and MusiQOL Scores at Week 12
Description: Correlation was assessed by using Pearson correlation coefficient. MSTCQ, HADS, FSS, PSQI and MusiQOL are described in the above endpoints. Following abbreviations used in the categories: Global side-effects (GLOBSE); description of pain (PAINDESCR).
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Number; unit: Correlation Coefficient
Arm/Group | Rebif Morning Administration | Rebif Evening Administration
Number analyzed (Participants) | 85 | 77
Correlation Coefficient
  Leptin and MSTCQ-ISR: Week 12: number analyzed (Participants) | 76 | 65
  Leptin and MSTCQ-ISR: Week 12 | 0.00595 | -0.10214
  Resistin and MSTCQ-ISR: Week 12: number analyzed (Participants) | 76 | 65
  Resistin and MSTCQ-ISR: Week 12 | -0.22380 | 0.04855
  Adiponectin and MSTCQ-ISR: Week 12: number analyzed (Participants) | 76 | 65
  Adiponectin and MSTCQ-ISR: Week 12 | -0.13365 | -0.14865
  Leptin and MSTCQ-GLOBSE: Week 12: number analyzed (Participants) | 85 | 76
  Leptin and MSTCQ-GLOBSE: Week 12 | 0.03121 | 0.21425
  Resistin and MSTCQ-GLOBSE: Week 12: number analyzed (Participants) | 85 | 76
  Resistin and MSTCQ-GLOBSE: Week 12 | 0.20285 | -0.12730
  Adiponectin and MSTCQ-GLOBSE: Week 12: number analyzed (Participants) | 85 | 76
  Adiponectin and MSTCQ-GLOBSE: Week 12 | 0.00169 | -0.06398
  Leptin and MSTCQ-benefits: Week 12: number analyzed (Participants) | 63 | 61
  Leptin and MSTCQ-benefits: Week 12 | 0.13023 | -0.10915
  Resistin and MSTCQ-benefits: Week 12: number analyzed (Participants) | 63 | 61
  Resistin and MSTCQ-benefits: Week 12 | -0.13544 | -0.15636
  Adiponectin and MSTCQ-benefits: Week 12: number analyzed (Participants) | 63 | 61
  Adiponectin and MSTCQ-benefits: Week 12 | 0.10726 | 0.04081
  Leptin and MSTCQ-PAINDESCR: Week 12: number analyzed (Participants) | 82 | 69
  Leptin and MSTCQ-PAINDESCR: Week 12 | 0.09118 | 0.01165
  Resistin and MSTCQ-PAINDESCR: Week 12: number analyzed (Participants) | 82 | 69
  Resistin and MSTCQ-PAINDESCR: Week 12 | -0.13918 | 0.04150
  Adiponectin and MSTCQ-PAINDESCR: Week12: number analyzed (Participants) | 82 | 69
  Adiponectin and MSTCQ-PAINDESCR: Week12 | 0.07093 | 0.01535
  Leptin and MSTCQ-VAS: Week 12: number analyzed (Participants) | 84 | 73
  Leptin and MSTCQ-VAS: Week 12 | 0.34840 | -0.01433
  Resistin and MSTCQ-VAS: Week 12: number analyzed (Participants) | 84 | 73
  Resistin and MSTCQ-VAS: Week 12 | -0.15231 | 0.16220
  Adiponectin and MSTCQ-VAS: Week 12: number analyzed (Participants) | 84 | 73
  Adiponectin and MSTCQ-VAS: Week 12 | -0.07840 | 0.02109
  Leptin and MSTCQ-pain rating: Week 12: number analyzed (Participants) | 85 | 75
  Leptin and MSTCQ-pain rating: Week 12 | 0.16675 | -0.14381
  Resistin and MSTCQ-pain rating: Week 12: number analyzed (Participants) | 85 | 75
  Resistin and MSTCQ-pain rating: Week 12 | -0.23531 | 0.12355
  Adiponectin and MSTCQ-pain rating: Week12: number analyzed (Participants) | 85 | 75
  Adiponectin and MSTCQ-pain rating: Week12 | -0.08060 | -0.08718
  Leptin and HADS-anxiety: Week 12: number analyzed (Participants) | 83 | 76
  Leptin and HADS-anxiety: Week 12 | 0.00754 | -0.06360
  Resistin and HADS-anxiety: Week 12: number analyzed (Participants) | 83 | 76
  Resistin and HADS-anxiety: Week 12 | 0.02447 | 0.07986
  Adiponectin and HADS-anxiety: Week 12: number analyzed (Participants) | 83 | 76
  Adiponectin and HADS-anxiety: Week 12 | 0.06295 | 0.08818
  Leptin and HADS-depression: Week 12: number analyzed (Participants) | 83 | 76
  Leptin and HADS-depression: Week 12 | 0.05226 | -0.14953
  Resistin and HADS-depression: Week 12: number analyzed (Participants) | 83 | 76
  Resistin and HADS-depression: Week 12 | 0.01970 | -0.04154
  Adiponectin and HADS-depression: Week 12: number analyzed (Participants) | 83 | 76
  Adiponectin and HADS-depression: Week 12 | 0.03228 | 0.19209
  Leptin and FSS: Week 12: number analyzed (Participants) | 81 | 77
  Leptin and FSS: Week 12 | 0.04256 | 0.14284
  Resistin and FSS: Week 12: number analyzed (Participants) | 81 | 77
  Resistin and FSS: Week 12 | -0.23755 | -0.10961
  Adiponectin and FSS: Week 12: number analyzed (Participants) | 81 | 77
  Adiponectin and FSS: Week 12 | -0.00326 | 0.03090
  Leptin and PSQI: Week 12: number analyzed (Participants) | 52 | 43
  Leptin and PSQI: Week 12 | 0.00873 | 0.00099
  Resistin and PSQI: Week 12: number analyzed (Participants) | 52 | 43
  Resistin and PSQI: Week 12 | -0.03765 | 0.12085
  Adiponectin and PSQI: Week 12: number analyzed (Participants) | 52 | 43
  Adiponectin and PSQI: Week 12 | 0.25795 | 0.24406
  Leptin and MusiQoL- Global: Week 12: number analyzed (Participants) | 74 | 64
  Leptin and MusiQoL- Global: Week 12 | -0.25650 | 0.17917
  Resistin and MusiQoL-Global: Week 12: number analyzed (Participants) | 74 | 64
  Resistin and MusiQoL-Global: Week 12 | 0.12190 | 0.21936
  Adiponectin and MusiQoL-Global: Week 12: number analyzed (Participants) | 74 | 64
  Adiponectin and MusiQoL-Global: Week 12 | 0.07152 | -0.05924

12. Secondary Outcome: Change From Baseline in Cytokines (Leptin and Resistin) Levels at Week 12
Description: Results are presented for cytokines: leptin and resistin.
Time Frame: Baseline and Week 12
Population: The Sub study Analysis Set (SSAS) included all subjects in the ITT who were enrolled in the sub study. Here, "Number of Subjects Analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Nanogram/milliliter (ng/mL)
Arm/Group | Rebif Morning Administration | Rebif Evening Administration
Number analyzed (Participants) | 8 | 7
Nanogram/milliliter (ng/mL)
  Leptin: Change at Week 12 | -2.7826 [-6.1880 to 0.6227] | -0.7936 [-4.4371 to 2.8499]
  Resistin: Change at Week 12 | -3.6628 [-5.3424 to -1.9831] | -5.8360 [-7.6339 to -4.0381]

13. Secondary Outcome: Change From Baseline in Cytokine (Adiponectin) Level at Week 12
Time Frame: Baseline and Week 12
Population: The SSAS included all subjects in the ITT who were enrolled in the sub study. Here, "Number of Subjects Analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: microgram per milliliter (mcg/mL)
Arm/Group | Rebif Morning Administration | Rebif Evening Administration
Number analyzed (Participants) | 8 | 7
microgram per milliliter (mcg/mL) | 2.7093 [-1.0663 to 6.4848] | 4.3574 [0.3174 to 8.3975]

14. Secondary Outcome: Change From Baseline in Hormone-Like Cytokine (Interleukin-6, 10 and 12) Levels at Week 12
Time Frame: Baseline and Week 12
Population: The SSAS included all subjects in the ITT who were enrolled in the sub study. Here, "Number of Subjects Analyzed" signifies those subjects who were evaluable for this outcome measure. Here "Number Analyzed" signifies those subjects who were evaluable for this outcome measure for specified category.
Measure: Least Squares Mean (95% Confidence Interval); unit: Pico gram/milliliter (pg/mL)
Arm/Group | Rebif Morning Administration | Rebif Evening Administration
Number analyzed (Participants) | 8 | 7
Pico gram/milliliter (pg/mL)
  Interleukin-6: Change at Week 12 | -0.5173 [-1.7940 to 0.7593] | -0.6970 [-2.0624 to 0.6683]
  Interleukin-10: Change at Week 12: number analyzed (Participants) | 5 | 3
  Interleukin-10: Change at Week 12 | -0.05819 [-0.5453 to 0.4290] | -0.6660 [-1.2999 to -0.03210]
  Interleukin-12: Change at Week 12: number analyzed (Participants) | 7 | 7
  Interleukin-12: Change at Week 12 | -0.3490 [-0.9115 to 0.2135] | -0.4384 [-0.9973 to 0.1204]

15. Secondary Outcome: Change From Baseline in Total Sleep Time (TST) and Rapid Eye Movement (REM) Sleep Time at Week 12
Description: Polysomnography (PSG) was performed for subjects who participated in the sub study. PSG is a multi-parametric test used in the study of sleep and as a diagnostic tool in sleep medicine. Total sleep time is the total of all REM and non-REM sleep in a sleep episode.
Time Frame: Baseline and Week 12
Population: as for outcome 14
Measure: Median (Full Range); unit: minutes
Arm/Group | Rebif Morning Administration | Rebif Evening Administration
Number analyzed (Participants) | 7 | 6
minutes
  Total Sleep Time: Change at Week 12 | 10.0 [-73.0 to 117.0] | 33.0 [-227.0 to 165.0]
  REM sleep: Change at Week 12: number analyzed (Participants) | 4 | 5
  REM sleep: Change at Week 12 | -3.0 [-207.0 to 9.0] | 6.0 [-67.0 to 288.0]

16. Secondary Outcome: Correlation Between Change From Baseline in Cytokines (Leptin, Resistin and Adiponectin) and Hormone-like Cytokine Levels (Interleukin-6, 10 and 12), and TST and REM Sleep Time at Week 12
Description: Correlations between change from baseline at Week 12 in TST or REM sleep and the area under the curve (AUC) calculated using the trapezoidal method for cytokine levels (i.e., leptin, resistin, adiponectin, Interleukin (IL)-12, IL 10, and IL 6) were analyzed using Pearson's correlation coefficient. Polysomnography (PSG) was performed for subjects who participated in the sub study.
Time Frame: Baseline and Week 12
Population: as for outcome 14
Measure: Number; unit: Correlation Coefficient
Arm/Group | Rebif Morning Administration | Rebif Evening Administration
Number analyzed (Participants) | 7 | 6
Correlation Coefficient
  AUC Leptin and TST: Week 12 | 0.10816 | 0.46984
  AUC Resistin and TST: Week 12 | -0.56278 | -0.05056
  AUC Adiponectin and TST: Week 12: number analyzed (Participants) | 7 | 5
  AUC Adiponectin and TST: Week 12 | 0.17402 | 0.58181
  AUC IL-12 and TST: Week 12: number analyzed (Participants) | 5 | 5
  AUC IL-12 and TST: Week 12 | -0.44328 | 0.24717
  AUC IL-10 and TST: Week 12: number analyzed (Participants) | 2 | 1
  AUC IL-10 and TST: Week 12 | 1.00000 | NA — Correlation Coefficient could not be estimated as there was only 1 subject analyzed for this arm at the specified time point.
  AUC IL-6 and TST: Week 12 | 0.18626 | -0.51662
  AUC Leptin and REM: Week 12: number analyzed (Participants) | 4 | 5
  AUC Leptin and REM: Week 12 | 0.99732 | 0.63155
  AUC Resistin and REM: Week 12: number analyzed (Participants) | 4 | 5
  AUC Resistin and REM: Week 12 | 0.22684 | -0.38234
  AUC Adiponectin and REM: Week 12: number analyzed (Participants) | 4 | 4
  AUC Adiponectin and REM: Week 12 | 0.98335 | -0.05732
  AUC IL-12 and REM: Week 12: number analyzed (Participants) | 2 | 4
  AUC IL-12 and REM: Week 12 | 1.00000 | -0.76606
  AUC IL-10 and REM: Week 12: number analyzed (Participants) | 2 | 1
  AUC IL-10 and REM: Week 12 | -1.00000 | NA — Correlation Coefficient could not be estimated as there was only 1 subject analyzed for this arm at the specified time point.
  AUC IL-6 and REM: Week 12: number analyzed (Participants) | 4 | 5
  AUC IL-6 and REM: Week 12 | 0.06269 | -0.34860

17. Secondary Outcome: Number of Subjects With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, TEAEs Leading to Death and TEAEs Leading to Discontinuation
Description: An adverse event (AE) was defined as any untoward medical occurrence in a subject which does not necessarily have a causal relationship with the treatment. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. The term TEAE is defined as AEs starting or worsening after the first intake of the study drug.
Time Frame: Baseline up to Week 12
Population: The Safety Analysis Set (SAF) included all subjects in the ITT who received at least 1 dose of the planned study treatment.
Measure: Number; unit: Subjects
Arm/Group | Rebif Morning Administration | Rebif Evening Administration
Number analyzed (Participants) | 104 | 96
Subjects
  TEAEs | 82 | 77
  Serious TEAEs | 1 | 2
  TEAEs Leading to Death | 0 | 0
  TEAE leading to Discontinuation | 6 | 3

ADVERSE EVENTS:
Time Frame: Baseline up to Week 12
Arm/Group | Rebif Morning Administration | Rebif Evening Administration
Serious Adverse Events (participants affected / at risk) | 1/104 | 2/96
Other Adverse Events (participants affected / at risk) | 77/104 | 70/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rebif Morning Administration (N=104) | Rebif Evening Administration (N=96)
Influenza Like Illness (General disorders) | 1 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rebif Morning Administration (N=104) | Rebif Evening Administration (N=96)
Nausea (Gastrointestinal disorders) | 10 | 2
Influenza Like Illness (General disorders) | 52 | 42
Pyrexia (General disorders) | 15 | 11
Injection Site Erythema (General disorders) | 14 | 8
Fatigue (General disorders) | 9 | 2
Asthenia (General disorders) | 7 | 4
Injection Site Pain (General disorders) | 5 | 5
Alanine Aminotransferase Increased (Investigations) | 4 | 7
Aspartate Aminotransferase Increased (Investigations) | 4 | 5
Transaminases Increased (Investigations) | 4 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 7
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4 | 6
Headache (Nervous system disorders) | 23 | 16
Multiple Sclerosis Relapse (Nervous system disorders) | 3 | 7
Insomnia (Psychiatric disorders) | 2 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other